CLINICAL TRIAL: NCT01943500
Title: Collection of Blood Specimens for Circulating Tumor Cell Analysis
Status: Completed | Type: Observational
Sponsor: Viatar LLC (Industry)
Collaborators: Commonwealth Hematology-Oncology, P.C. (Unknown)
Responsible Party: Sponsor
Other Study IDs: T30-0001
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer
Keywords: Breast cancer; Prostate cancer; Colorectal cancer; Circulating tumor cell (CTC)
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer or no prior history of cancer: Confirmed patients with breast, prostate, or colorectal cancer (OR) subjects with no prior history of cancer

SUMMARY:
Objective: To test the sensitivity of a proprietary novel filtration device designed to capture and concentrate circulating tumor cells (CTCs).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Written informed consent obtained
* Confirmed diagnosis of stage 2-4 breast, prostate, or colorectal cancer, (OR) no prior history of cancer
* Stage 2-4 treatment naive, metastatic, secondary, and recurrent cancer patients
* Able to undergo blood collection prior to initiation of chemotherapy treatment, (OR) able to provide blood sample if subject is a non-cancer control subject

Exclusion Criteria:

* Patients unable to understand the research protocol and/or provide informed consent.
* Patients with known immunodeficiency, or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed patients with stage II-IV breast, prostate, or colorectal cancer, (Or) subjects with no prior history of cancer.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2014-01-28 (Actual); Study Completion 2016-08-26 (Actual)

PRIMARY OUTCOMES:
The number of circulating tumor cells (CTCs) per milliliter of whole blood. Reported unit of measure will be the number of CTCs/milliliter. | Analysis will be performed within 96 hours following blood sample collection
  Blood samples will be collected from study subjects and analyzed for the number of circulating tumor cells (CTCs) within 96 hours of blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro M Sanz-Altamira, MD, PhD, Principal Investigator — Commonwealth Hematology-Oncology, P.C.
Locations (1):
- Commonwealth Hematology-Oncology, P.C., Lawrence, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No